CLINICAL TRIAL: NCT00390234
Title: A Phase II Study of VEGF-Trap in Recurrent or Metastatic Gynecologic Soft-Tissue Sarcomas
Brief Title: Ziv-aflibercept in Treating Patients With Locally Advanced, Unresectable, or Metastatic Gynecologic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00177; PHL-051 (Other Grant/Funding Number: N01CM62209); CDR0000508798 (Other Grant/Funding Number: N01CM62209); N01CM62209 (NIH); N01CM62203 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2013-05

CONDITIONS: Fallopian Tube Cancer; Female Reproductive Cancer; Ovarian Carcinosarcoma; Ovarian Sarcoma; Recurrent Ovarian Epithelial Cancer; Recurrent Uterine Sarcoma; Stage III Ovarian Epithelial Cancer; Stage III Uterine Sarcoma; Stage IV Ovarian Epithelial Cancer; Stage IV Uterine Sarcoma; Uterine Carcinosarcoma; Uterine Leiomyosarcoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ziv-aflibercept) (Experimental): Patients receive ziv-aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ziv-aflibercept

INTERVENTIONS:
Drug: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap

SUMMARY:
This phase II trial is studying how well ziv-aflibercept works in treating patients with locally advanced, unresectable or metastatic gynecologic soft tissue sarcoma. Ziv-aflibercept may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response of recurrent or metastatic gynecologic soft-tissue sarcomas to VEGF-Trap (ziv-aflibercept).

II. To assess the incidence of disease stabilization, as measured by 6-month progression-free survival, in patients with recurrent or metastatic gynecologic soft-tissue sarcomas treated with VEGF-Trap.

SECONDARY OBJECTIVES:

I. To assess time-to-progression and overall survival in patients with recurrent or metastatic gynecologic soft-tissue sarcoma treated with VEGF-Trap.

* As of 24 October 2012, overall survival follow-up is to be discontinued for the one remaining patient on long term follow-up, who has been off protocol therapy for at least 3 years. Time to progression and median survival times have been based on the currently available data.

II. To assess the toxicity associated with VEGF-Trap in patients with recurrent or metastatic gynecologic soft-tissue sarcoma.

III. To characterize the population pharmacokinetics of VEGF-Trap and to explore for demographic and clinical covariates

OUTLINE: This is an open-label, multicenter study.

Patients are stratified according to histology (uterine leiomyosarcoma vs malignant mixed mullerian tumor/carcinosarcoma). Patients receive ziv-aflibercept over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood collection at baseline, every 8 weeks during treatment, and 60 days after completion of study treatment for population pharmacokinetic analysis using enzyme-linked immunosorbent assay (ELISA).

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed soft tissue sarcoma of gynecologic tract including 1 of the following subtypes: uterine leiomyosarcoma, malignant mixed mullerian tumor/carcinosarcoma, disease originating in ovary/fallopian tube allowed
* Locally advanced/unresectable/metastatic disease
* Previously treated disease must have radiographic/clinical evidence of PD
* Measurable disease-at least 1 lesion in at least 1 dimension (longest diameter) as >=20mm with conventional techniques or as >=10mm with spiral CT scan
* Indicator lesions may not have been previously treated with surgery/radiotherapy/radiofrequency ablation unless PD has been confirmed
* ECOG PS 0-2 OR Karnofsky PS 60-100%
* Life expectancy>=3 months
* WBC>=3,000/mm^3
* Absolute neutrophil count>=1,500/mm^3
* Platelet count>=75,000/mm^3
* Bilirubin=<1.5xULN
* AST and ALT=<3xULN
* INR=<1.5 (unless on warfarin)
* Creatinine=<1.5xULN OR creatinine clearance>=60 mL/min
* Urine protein<1+ by dipstick OR 24-hour urine protein<500 mg OR urine protein:creatinine ratio<1
* Not pregnant/nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥6 months after treatment - No other active malignancy within past 5 years except adequately treated cervical carcinoma in situ/nonmelanoma skin cancer
* No known hypersensitivity to Chinese hamster ovary cell products/other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical/biological composition to study agents
* No serious/nonhealing wound/ulcer/bone fracture
* No abdominal fistula/gastrointestinal perforation/bowel obstruction/intraabdominal abscess within past 28 days
* No significant traumatic injuries within past 28 days
* No evidence of bleeding diathesis/coagulopathy
* No uncontrolled intercurrent illness including but not limited to: Ongoing/active infection, psychiatric illness or social situations that would preclude study compliance
* <=2 prior cytotoxic chemotherapy regimen for recurrent, locally advanced or metastatic disease
* Recovered from prior therapy
* No prior antiangiogenic agent

Exclusion Criteria:

* < 4weeks since prior chemotherapy (<6 weeks for nitrosoureas/carmustine/mitomycin C), prior investigational treatment, radiotherapy and major surgery/open biopsy
* 1 week since prior core biopsy
* 1 month since prior thrombolytic agents
* Concurrent full-dose anticoagulants with INR>1.5 allowed if: In-range INR (usually between 2-3) on stable dose of oral anticoagulant or low molecular weight heparin,
* OR; For patients on warfarin, the upper target for INR is ≤3 No active bleeding/pathological condition that carries a high risk of bleeding (e.g. tumor invading major vessels/known varices)
* No evidence of CNS disease including primary brain tumor/brain metastasis
* No other concurrent investigational agents - No concurrent major surgery
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Clinically significant cardiovascular disease including:

  * Cerebrovascular accident within past 6 months,
  * Uncontrolled hypertension defined as BP>150/100mmHg OR systolic BP>180mmHg if diastolic BP<90 mmHg, on ≥2 repeated determinations on separate days within past 3 months,
* OR; Antihypertensive medications allowed as long as dose and number of antihypertensive medications have not increased within past 2 weeks, Myocardial infarction, coronary artery bypass graft, or unstable angina within past 6 months, OR;
* OR; NYHA class III-IV congestive heart failure, serious cardiac arrhythmia requiring medication, or unstable angina pectoris within past 6 months, Clinically significant peripheral vascular disease within past 6 months
* OR; pulmonary embolism, deep vein thrombosis, or other thromboembolic event within past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (16):
- United States (8):
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Peoria Gynecologic Oncology, Peoria, Illinois
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Fox Chase Cancer Center, Rockledge, Pennsylvania
- Canada (8):
  - Vancouver General Hospital, Vancouver, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ziv-aflibercept): Patients receive ziv-aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Ziv-aflibercept)
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 78]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
  Canada | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Evaluated According to the RECIST Criteria
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 63
participants | 0

2. Primary Outcome: Incidence of Disease Stabilization, as Measured by Progression-free Survival at 6 Months (Leiomyosaroma Group)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 40
months | 0.17 [0.06 to 0.32]

3. Secondary Outcome: Survival (Leiomyosarcoma Group)
Description: Survival statistics will be estimated using the Kaplan-Meier method. Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. 95% confidence intervals will be provided for estimates of interest where possible.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 40
months | 18.1 [8.5 to NA] — Value not reached

4. Primary Outcome: Incidence of Disease Stabilization, as Measured by Progression-free Survival at 6 Months (Carcinosarcoma Group)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 22
months | 1.6 [1.1 to 1.7]

5. Secondary Outcome: Survival (Carcinosarcoma Group)
Description: as for outcome 3
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 22
months | 3.2 [1.4 to NA] — Value not reached

ADVERSE EVENTS:
Arm/Group | Treatment (Ziv-aflibercept)
Serious Adverse Events (participants affected / at risk) | 29/63
Other Adverse Events (participants affected / at risk) | 47/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ziv-aflibercept) (N=63)
Anemia (Blood and lymphatic system disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Creatinine increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Death NOS (General disorders) | 4
Hypotension (Vascular disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Hypertension (Vascular disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Edema limbs (General disorders) | 1
Headache (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Lymphocyte count decreased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 4
Small intestinal perforation (Gastrointestinal disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 1
Urinary tract infection (Infections and infestations) | 1
Fatigue (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vitreous hemorrhage (Eye disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ziv-aflibercept) (N=63)
Fatigue (General disorders) | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less